CLINICAL TRIAL: NCT03766308
Title: The Clinical Study of the Effect of Highland Barley Diet on Blood Glucose in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuefeng Yu (Other)
Responsible Party: Sponsor-Investigator, Xuefeng Yu, Director of Department of Endocrinology, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJ-NFM-0001
Record Dates: First submitted 2017-10-29; First posted 2018-12-06 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: highland barley diet
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Highland barley diet (Experimental): highland barley diet(20g, thrice-daily) +Metformin sustained-release tablets(500mg, thrice-daily)
  Interventions: Dietary Supplement: Highland Barley Diet
- ADA diet (Active Comparator): ADA diet + Metformin sustained-release tablets(500mg, thrice-daily)
  Interventions: Dietary Supplement: ADA diet

INTERVENTIONS:
Dietary Supplement: Highland Barley Diet — Highland Barley Diet
  Arms: Highland barley diet
Dietary Supplement: ADA diet — ADA diet
  Arms: ADA diet

SUMMARY:
The clinical study of the effect of highland barley diet on blood glucose in patients with type 2 diabetes mellitus

DETAILED DESCRIPTION:
The clinical study of the effect of highland barley diet on blood glucose in patients with type 2 diabetes mellitus.

Approximately 40 patients will be enrolled in the study from China and randomized in a 1:1 ratio to one of the 2 treatment arms: highland barley diet + metformin; or +common diet metformin.

Study treatment will continue for 12 weeks. The primary efficacy measure is the change in HbA1c at 12 weeks. The study consists of 3 periods: a 1-week screening (period A), a 4-week run-in period (period B) and a 12-week treatment period (period C).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Type 2 diabetic patients （new diagnose ）
3. HbA1c ≥7.0 % and < 9.0 % (HbA1c > 7.0 % and ≤ 8.0% at randomization)
4. Men and women (non-pregnant and using a medically approved birth-control method) aged ≥ 18 and ≤ 70 years
5. BMI ≥ 23 and ≤ 35 kg/m2

Exclusion Criteria:

1. Type 1 diabetes or other specific types of diabetes
2. Pregnancy, preparation for pregnancy, lactation and women of child-bearing age incapable of effective contraception methods
3. Uncooperative subject because of various reasons
4. Abnormal liver function, glutamic-pyruvic transaminase (ALT) and glutamic-oxaloacetic transaminase (AST) > twice the upper limits of normal
5. Impairment of renal function, serum creatinine: ≥ 133mmol/L for female，≥ 135mmol/L for male
6. Serious chronic gastrointestinal diseases
7. Edema
8. Serious heart diseases, such as cardiac insufficiency (level III or more according to NYHA), acute coronary syndrome and old myocardial infraction
9. Blood pressure: Systolic blood pressure (SBP) ≥ 180mmHg and/or diastolic blood pressure (DBP) ≥ 110mmHg
10. White blood count (WBC) < 4.0×109/L or platelet count (PLT) < 90×109/L，or definite anemia (Hb：< 120g/L for male, < 110g/L for female), or other hematological diseases
11. Endocrine system diseases, such as hyperthyroidism and hypercortisolism
12. Experimental drug allergy or frequent hypoglycemia
13. Psychiatric disorders, drug or other substance abuse
14. Diabetic ketoacidosis and hyperosmolar nonketotic coma requiring insulin therapy
15. Stressful situations such as surgery, serious trauma and so on
16. Chronic hypoxic diseases such as pulmonary emphysema and pulmonary heart disease
17. Combined use of drugs effecting glucose metabolism such as glucocorticoid Tumor, especially bladder tumor and/or family history of bladder tumor and/or long-term hematuria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
HbA1c | from baseline to 12-week endpoint
  In the newly diagnosed type 2 diabetic patients, the absolute value of glycosylated hemoglobin from baseline to 12-week endpoints was compared between groups in the qingke diet group and the normal diet group.

SECONDARY OUTCOMES:
The percentage of participants who achieved HbA1c ≤ 6.5% and < 7% | 12 weeks
  The percentage of participants who achieved HbA1c ≤ 6.5% and < 7%
blood glucose | 6 weeks and 12weeks
  Fasting blood glucose
Postprandial Blood Glucose | 6 weeks and 12weeks
  Postprandial blood glucose
7 point self-monitoring blood sugar | from baseline to 6 and 12 weeks
  7 point self-monitoring blood sugar
blood lipid | from baseline to 6 and 12 weeks
  blood lipid
uric acid | from baseline to 6 and 12 weeks
  uric acid
Insulin resistance index | 0weeks and 12weeks
  Insulin resistance index
Beta cell function index of islet | 0weeks and 12weeks
  Beta cell function index of islet
Change in body weight | from baseline to 12 weeks
  Change in body weight
Change in Waist circumference | from baseline to 12 weeks
  Change in Waist circumference

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and technology, Wuhan, Hubei, China